CLINICAL TRIAL: NCT04207671
Title: Omission of Chest Tube Versus Improved Drainage Strategy in Patients With Lung Wedge Resection: A Prospective Randomized Trial
Brief Title: Improved Drainage Strategy for Patients With Lung Wedge Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Porfessor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TBL-2
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Drainage
Keywords: Tubeless; Wedge resection; Improved drainage strategy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omission of chest tube (Other): After wedge resection and the air-leak test, patients will receive complete omission of chest tube and directly close the incision.
  Interventions: Procedure: Complete omission of chest tube
- Improved drainage strategy (Experimental): After wedge resection and the air-leak test, patients willreceive a two-lumen central venous catheterization along the midclavicular line, second intercostal space for remedial gas-removal.
  Interventions: Procedure: Improved drainage strategy

INTERVENTIONS:
Procedure: Complete omission of chest tube — No chest tube implacement
  Arms: Omission of chest tube
Procedure: Improved drainage strategy — A two-lumen central venous catheterization along the midclavicular line, second intercostal space for remedial gas-remove
  Arms: Improved drainage strategy

SUMMARY:
This study evaluates the viability and safety of two-lumen catheterization versus complete omission of chest tube in patients with lung wedge resection. Half of participants will receive complete omission of chest tube, while the other half will receive a two-lumen central venous catheterization along the midclavicular line, second intercostal space for remedial gas-remove.

DETAILED DESCRIPTION:
With the development of video-assisted thoracoscopic surgery (VATS) techniques, minimally invasive thoracic surgery has evolved considerably over the last three decades. The concept of "tubeless" involves non-intubated anesthesia with spontaneous ventilation and no chest tube placement. Chest tube placement always causes pain, and its duration is known to be one of the most important factors influencing hospital stay and costs. Early tube removal allows patients to breathe deeply with less pain, which leads to more compliance with chest physiotherapy, as demonstrated by a concomitant improvement in patients' ventilatory function. Hence, more and more experienced surgeons choose the omission of chest tube placement after lung wedge resection. However, based on previous retrospective studies, residual pneumothorax was noted in about 10% cases, and some of them need re-intervention. Hence, the investigators designed a intra-operative two-lumen catheterization as improved drainage strategy. Therefore, this study evaluates the viability and safety of two-lumen catheterization versus omission of chest tube placement in patients with lung wedge resection.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative radiology revealed solitary peripheral pulmonary nodule, with both size and depth less than 3 cm
2. Lung wedge resection for tumor biopsy to elucidate drug resistant mechanism or confirm diagnosis

Exclusion Criteria:

1. Previous ipsilateral thoracic surgery or extensive adhesion
2. Preoperative radiology revealed pneumonia or atelectasis
3. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
4. Bleeding tendency or anticoagulant use
5. Pregnancy or breast feeding
6. Patient who can not sign permit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of massive pneumothorax on day 1 after surgery | 1 day
  To evaluate the incidence rate of pneumothorax (a pneumothorax greater than 2.0 cm on X-ray)

SECONDARY OUTCOMES:
Pain score on day 1 after surgery | 1 day
  To evaluate the pain score via numerical rating scale on day 1 after surgery. An 11-point numeric scale (NRS 11) with 0 representing no pain and 10 representing worst pain imaginable.
Length of post-operative hospital stay | 1 week
  To evaluate the length of post-operative hospital stay.
Postoperative pulmonary function recovery | 1 month
  To evaluate the postoperative cardiopulmonary function recovery via 6-minute walk test in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Song Dong, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang JT, Tang YC, Lin JT, Dong S, Nie Q, Jiang BY, Yan HH, Wen ZW, Wu Y, Yang XN, Wu YL, Zhong WZ. Prophylactic air-extraction strategy after thoracoscopic wedge resection. Thorac Cancer. 2018 Nov;9(11):1406-1412. doi: 10.1111/1759-7714.12850. Epub 2018 Sep 6. PMID 30187689